CLINICAL TRIAL: NCT01873222
Title: OPtical Frequency Domain Imaging vs. INtravascular Ultrasound in Percutaneous Coronary InterventiON - OPINION Imaging
Brief Title: OPtical Frequency Domain Imaging Versus INtravascular Ultrasound in Percutaneous Coronary InterventiON - OPINION Imaging
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Wakayama Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TRICVD1311; UMIN000010581 (Registry Identifier: UMIN Clinical Trial Registry)
Record Dates: First submitted 2013-05-27; First posted 2013-06-10 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Percutaneous Coronary Intervention; Optical Frequency Domain Imaging; Intravascular Ultrasound
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OFDI-guided PCI & IVUS (Experimental): * Assessment by IVUS at post-PCI
  * Assessment by OFDI at a 8-month follow-up
  Interventions: Device: OFDI-guided PCI & IVUS
- IVUS-guided PCI & OFDI (Active Comparator): * Assessment by OFDI at post-PCI
  * Assessment by OFDI at a 8-month follow-up
  Interventions: Device: IVUS-guided PCI & OFDI

INTERVENTIONS:
Device: OFDI-guided PCI & IVUS — * Assessment by IVUS at post-PCI
  * Assessment by OFDI at a 8-month follow-up
  Other Names: OFDI; LUNAWAVE; Biolimus A9-eluting stent (Nobori stent)
  Arms: OFDI-guided PCI & IVUS
Device: IVUS-guided PCI & OFDI — * Assessment by OFDI at post-PCI
  * Assessment by OFDI at a 8-month follow-up
  Other Names: VISIWAVE; ViewIT; Biolimus A9-eluting stent (Nobori stent)
  Arms: IVUS-guided PCI & OFDI

SUMMARY:
This study is the sub-study of OPINION Trial. (UMIN000010580) The aim of this study is to evaluate how Optical frequency domain imaging (OFDI) or Intravascular Ultrasound (IVUS) imaging technology influence to the Percutaneous Coronary Intervention (PCI) strategy.

DETAILED DESCRIPTION:
Optical frequency domain imaging (OFDI) is a novel, high resolution intravascular imaging modality. Intravascular ultrasound (IVUS) is a widely used conventional imaging modality for achieving optimal stent deployment.

This study is the sub-study of OPINION Trial. (UMIN000010580) The aim of this study is to evaluate how OFDI or IVUS imaging technology influence to the Percutaneous Coronary Intervention (PCI) strategy.

We will enroll the first 100 patients who have enrolled in the main-study of OPINION trial.(UMIN000010580). We will assess lesions by the other device in addition to the assigned device in the main study at the time of post-PCI.

We will then assess lesions by OFDI at a 8-month follo-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients participating in the OPINION Trial
* Patients who has provided written informed consent

Exclusion Criteria:

* Ineligible patients according to the investigator's judgment
* Inability or unwillingness to perform required follow up procedures

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2013-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Minimum stent area by OFDI | at just after the PCI
  The investigators will assess "Minimum stent area" by OFDI at post-PCI.
Frequency of malapposed struts | at just after the PCI
  The investigators will assess "Frequency of malapposed struts" by OFDI at post-PCI.
Dissection | at just after the PCI
  The investigators will assess "Dissection" by OFDI at post-PCI.
Minimum stent area by IVUS | at just after the PCI
  The investigators will assess "Minimum stent area" by IVUS at post-PCI.
Frequency of uncovered struts | 8 months after PCI
  The investigators will assess "Frequency of uncovered struts" by OFDI at 8 months after PCI.
Minimum lumen area | 8-month follow-up after PCI
  The investigators will assess "Minimum lumen area by OFDI at 8 months after PCI.

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Akasaka, MD, PhD, Principal Investigator — Wakayama Medical University
Locations (1):
- Wakayama Medical University, Wakayama, Wakayama, Japan

REFERENCES:
- [Derived] Otake H, Kubo T, Takahashi H, Shinke T, Okamura T, Hibi K, Nakazawa G, Morino Y, Shite J, Fusazaki T, Kozuma K, Ioji T, Kaneda H, Akasaka T; OPINION Investigators. Optical Frequency Domain Imaging Versus Intravascular Ultrasound in Percutaneous Coronary Intervention (OPINION Trial): Results From the OPINION Imaging Study. JACC Cardiovasc Imaging. 2018 Jan;11(1):111-123. doi: 10.1016/j.jcmg.2017.06.021. Epub 2017 Oct 5. PMID 28917678